CLINICAL TRIAL: NCT02146248
Title: Tubal Patency During the Menstrual Cycle and During Treatment With Hormonal Contraceptives: a Pilot Study in Women
Brief Title: HSG and Tubal Patency Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Jensen (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Jensen, Dr. Jeffrey Jensen, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OHSU IRB 10103
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Tubal Patency
Keywords: hysterosalpingography, DMPA, combined oral contraceptive, tubal patency
MeSH Terms: interventions — Contraceptives, Oral, Combined; Contraceptives, Oral; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSG Studies (Experimental): Women will be given combined oral contraceptives and Depo-medroxyprogesterone acetate (DepoProvera®).
  2 HSG studies will be done prior to hormonal treatment, 1 after the pill treatment, and depending on whether the tubes appear patent, 1 more after the depoProvera treatment, and a final HSG after another 2 weeks on the pill.
  Interventions: Drug: combined oral contraceptive; Drug: DepoProvera

INTERVENTIONS:
Drug: combined oral contraceptive — combined oral contraceptive pill will be dosed continuously for 30 days without cycle interruption
  Other Names: pill, birth control pill, COC
Drug: DepoProvera — injectable hormonal contraceptive
  Other Names: Depo-medroxyprogesterone acetate, DMPA

SUMMARY:
The investigators' research group is working to develop a highly effective, low cost non-surgical method of permanent contraception for women. To support this goal, we need to know more about the normal fallopian tube (tube that passes the egg from the ovary into the womb). The purpose of this study is to learn about how menstrual cycles and hormonal contraceptives affect tubal patency. Normally there is an opening between the tube and uterus to permit the flow of fluid and cells. If this opening is blocked, this can result in infertility. Tubal patency is when a woman's fallopian tubes are not blocked. Tubal patency is determined by an x-ray test called a hystero-(uterus)salpingo-(fallopian tube)graphy (HSG). HSG is a standard radiological imaging study that is used to determine if the fallopian tubes are open and free of disease. It is commonly done in women with an infertility diagnosis. The investigators usually do this test in the first 10 days of the menstrual cycle. Sometimes the tubes will appear to be blocked on the HSG when they are actually open. The timing of the HSG study during the menstrual cycle, or the use of hormonal contraception may make a difference in whether the tubes appear blocked on the HSG when they are actually patent.

The results of the HSG test provide a good model for how our nonsurgical permanent contraception method might work. The investigators think that if the tubes are not patent, that our treatment will not work as well. Therefore, in this study we want to learn if menstrual cycle timing or current hormonal contraception use will affect the patency of the tubes as assessed by the HSG. The investigators want to examine the same women to see if tubal patency is changes during the menstrual cycle and during the use of a birth control pill and the birth control shot.

ELIGIBILITY:
Inclusion Criteria:

i. Women between 18 and 40 years old ii. In good health, with regular menstrual cycles that occur 24 - 37 days iii. No current use of hormonal contraception or an intrauterine device and having had at least one complete menstrual cycle since having stopped hormonal contraception before starting the treatment.

iv. Have a negative urine pregnancy test at the admission visit. v. Have a negative chlamydia test at the admission visit. vi. Not be at risk for pregnancy. They will be consistently using a non-hormonal contraception method, have a surgically sterile male partner with a vasectomy, be abstinent, or be in a same-sex relationship from the screening visit through the first study cycle. After starting the combined OC (see Visit 4 below), use of a non-hormonal method is no longer required.

vii. In the opinion of the investigator, willing and able to follow all study requirements, including use of the approved study medications (doxycycline, oral contraceptive and DMPA).

viii. Understand and sign an IRB approved inform consent form prior to screening activities.

ix. Will have diastolic blood pressure (BP) ≤85 mm Hg and systolic BP ≤145 mm Hg after 5 minutes in sitting position.

x. Agree not to participate in any other clinical trials during the course of this study.

Exclusion Criteria:

* i. Women with menstrual cycle length of less than 24 or more than 37 days; or with spontaneous irregular menstrual cycle length with intra-individual variations of more than 5 days ii. Currently pregnant as confirmed by positive high-sensitivity urine pregnancy test iii. Women planning pregnancy within their months of study participation iv. Currently breast-feeding or within 30 days of discontinuing breast feeding v. Current use of a hormonal IUD, or other hormonal contraception (including oral contraceptives, contraceptive vaginal rings, contraceptive patches, or contraceptive implants) within 30 days prior to screening. NOTE: Discontinuation of hormonal contraception or removal of implanted hormonal contraceptives must have been for personal reasons unrelated to the purpose of enrollment in this study.

vi. Undiagnosed abnormal genital bleeding vii. Known hypersensitivity to radio-opaque contrast, doxycycline, levonorgestrel, ethinyl estradiol or depo-medroxyprogesterone acetate. The active ingredients in the approved medications used in the study.

viii. Anomalies in the clinical exam or history done at screening visit recognized as clinically significant by the investigator.

ix. Unable to pass a uterine sound at the screening examination. x. A positive test for chlamydia at screening, or a history of a positive test within the last 6 months.

xi. A clinically significant Pap test abnormality, as managed by current local or national guidelines that would require treatment over the next 6 months.

xii. Invasive cancer (past history of any carcinoma or sarcoma, except non-melanoma skin cancer) xiii. Body mass index (BMI) >35. xiv. Current use of a non-hormone containing (copper) intrauterine device (IUD). NOTE: Removal of an IUD must have been for personal reasons unrelated to the purpose of enrollment in this study.

xv. Smoking if > age 35. xvi. Personal history of venous or arterial thrombosis or embolism, or family history in a first-degree relative <55 years of age suggesting familial defect in blood coagulation system, which in the opinion of the principal investigator, suggests use of a hormonal contraceptive could pose a significant risk.

xvii. Cerebrovascular or cardiovascular disease. xviii. History of retinal vascular lesions, unexplained partial or complete loss of vision.

xix. Headaches with focal neurological symptoms. xx. History of cholestatic jaundice of pregnancy or jaundice with prior steroid use.

xxi. Use of liver enzyme inducers on a regular basis. xxii. History of involuntary infertility, pelvic inflammatory disease (not followed by a normal pregnancy), or known gynecologic conditions or surgery that could affect tubal patency (e.g. tubal adhesions, endometriosis, hydrosalpinx, salpingectomy, hysterectomy, oophorectomy).

xxiii. History of a prior HSG showing tubal occlusion on one or both sides.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jensen, MD MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: Women's Health Research Unit Website — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 subjects were screened, and 11 signed consent and enrolled. One dropped out prior to the first HSG, and10 completed the 2 natural cycle HSG, 9 completed the COC HSG, 7 the DMPA HSG, and one a final post DMPA HSG after restarting COCs
Groups:
- HSG Studies: Women will be given combined oral contraceptives and Depo-medroxyprogesterone acetate (DepoProvera®).
  2 HSG studies will be done prior to hormonal treatment, 1 after the pill treatment, and depending on whether the tubes appear patent, 1 more after the depoProvera treatment, and a final HSG after another 2 weeks on the pill.
  Combined oral contraceptive: combined oral contraceptive pill will be dosed continuously for 30 days without cycle interruption
  DepoProvera: injectable hormonal contraceptive
Period: Overall Study
Arm/Group | HSG Studies
Started | 11
Enrolled | 11
Uterine Sounding | 11 (one subject dropped out after uterine sound before HSG #1)
HSG 1 | 10
HSG 2 | 10
HSG 3 | 9
HSG 4 | 7
HSG 5 | 1
Completed | 9
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | HSG Studies
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Nulligravid [Count of Participants; unit: Participants] | 6
One or more births [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bilateral Tubal Patency as Assessed by HSG-follicular
Description: Assessment of patency at follicular phase exam
Time Frame: follicular phase HSG
Measure: Count of Participants; unit: Participants
Arm/Group | Follicular Phase HSG
Number analyzed (Participants) | 10
Participants
  bilateral patent | 9
  blocked | 1
Statistical Analysis 1: Comparison: Follicular Phase HSG; McNemar paired. Hypothesis is no change in tubal patency status. All subjects know to have bilateral patency in one of the exams during natural cycle; Test type: Superiority or Other; p = 0.4795, McNemar — The two-tailed P value equals 0.4795

2. Primary Outcome: Number of Participants With Bilateral Tubal Patency as Assessed by HSG - Luteal
Description: Assessment of patency at luteal phase exam
Time Frame: luteal phase HSG
Measure: Count of Participants; unit: Participants
Groups:
- Tubal Patency Change: Change in tubal patency after OC treatment
Arm/Group | Tubal Patency Change
Number analyzed (Participants) | 10
Participants
  bilateral tubal patency | 10
  blocked | 0

3. Other Pre Specified Outcome: Number of Participants With Bilateral Tubal Patency as Assessed by HSG - OC HSG
Description: HSG during OC treatment
Time Frame: HSG on OC
Measure: Count of Participants; unit: Participants
Groups:
- HSG 3: OC HSG
Arm/Group | HSG 3
Number analyzed (Participants) | 9
Participants
  bilateral tubal patency | 7
  blocked | 2

4. Other Pre Specified Outcome: Number of Participants With Bilateral Tubal Patency as Assessed by HSG - DMPA HSG
Description: HSG during DMPA treatment
Time Frame: HSG on DMPA
Measure: Count of Participants; unit: Participants
Groups:
- HSG 4: DMPA HSG
Arm/Group | HSG 4
Number analyzed (Participants) | 7
Participants
  bilateral patubal patency | 6
  blocked | 1

5. Other Pre Specified Outcome: Number of Participants With Bilateral Tubal Patency as Assessed by HSG -- Post DMPA Add Back COC HSG
Time Frame: HSG on OC after DMPA
Measure: Count of Participants; unit: Participants
Groups:
- HSG 5: post DMPA OC HSG
Arm/Group | HSG 5
Number analyzed (Participants) | 1
Participants
  bilateral patent | 1
  blocked | 0

ADVERSE EVENTS:
Time Frame: May 2014 - Feb 2015
Arm/Group | HSG Studies
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSG Studies (N=10)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a descriptive pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No